CLINICAL TRIAL: NCT05262543
Title: Redictive Risk Factors of Conversion Into Idiopathic RBD. Italian Study [FAttori di Rischio PREdittivi di Conversione Nell'RBD Idiopatico. STudio ItalianO
Brief Title: PREdictive Risk Factors of Conversion Into Idiopathic RBD. Italian Study
Acronym: FARPRESTO
Status: Recruiting | Type: Observational
Sponsor: University of Cagliari (Other)
Collaborators: University of Bologna (Other); University of Genova (Other); University of Pavia (Other); Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Monica Puligheddu, Professor of Neurology, University of Cagliari
Other Study IDs: FarPresto01
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: REM Sleep Behavior Disorder
Keywords: atonia; neurodegeneration
MeSH Terms: conditions — REM Sleep Behavior Disorder; Nerve Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
REM Sleep Behavior Disorder (RBD) is a REM sleep parasomnia first described in 1986 and characterized by the loss of physiological muscle atonia typical of REM sleep and by the presence of abnormal, sometimes violent, motor activity often related to dream content The observed motor behaviors are often associated to vivid dreams, characterized by an aggressive-defensive content, even if pleasant dreams have been described, resulting in non-violent behaviors. Diagnosis of RBD requires video-polysomnographic recording (vPSG) at a Sleep Center, essential to identify and quantify the complete or intermittent loss of physiological muscle atonia during REM sleep (REM sleep without atonia, RSWA) and record any related motor behaviors. The exact prevalence of RBD in the general population is not known and it seems underrated, but is estimated to be 0.3-1.15%. RBD is defined as idiopathic or isolated (iRBD) when it is not associated with other neurological diseases. The so-called symptomatic RBD, on the other hand, can occur in association with neurodegenerative diseases of the spectrum of alpha-synucleinopathies which include Parkinson's Disease (PD), Multiple System Atrophy (AMS), and Lewy Body Dementia (DLB). In recent years, several follow-up studies on large cohorts of iRBD patients have shown that the idiopathic form evolves towards a symptomatic form in most cases. More precisely, the risk of developing an alpha-synucleinopathies increases over time, with a conversion rate of up to 90% in some studies at 14 years. RBD represents an early marker of neurodegeneration, like a unique open window on the initial, pre-symptomatic phase of alpha-synucleinopathies, which could allow the use of neuroprotective therapies, as soon as they are available. Several longitudinal studies indicated older age, presence of hyposmia, abnormal color vision, minimal extrapyramidal motor signs, mild cognitive impairment, autonomic disturbances, and severity of loss of RSWA as risk factors for neurodegeneration. However, most studies investigated biomarkers separately, with retrospective study designs, in small cohorts or without a rigorous harmonization between centers in the case of multicenter studies.

To date, however, there is no reliable pool of biomarkers that predict the phenoconversion into α-synucleinopathy, the timing in which this can occur, and the phenotype of α-synucleinopathy. Furthermore, despite clinical and research evidence suggesting that iRBD is a heterogeneous disorder little attention was paid to different iRBD phenotypes and currently, there are no relevant data on the impact of iRBD on quality of life.

Actually, through neural network analysis approaches, it is possible to find out complex correlations between data from different sources (i.e., clinical examinations, questionnaires, biological data, imaging and neurophysiological techniques, etc.) and to identify subgroups of patients sharing the same substantial characteristics. Identifying different iRBD phenotypes through established as well as innovative biomarkers and standardized measures of wellbeing is crucial to better understanding alpha-synucleinopathies, developing targeted interventions, and reducing the disease burden.

To this aim, clinical, biological, neurophysiological, neuropsychological and imaging biomarkers need to be prospectively collected, according to standardized and harmonized procedures. This would significantly increase our understanding of the physiopathological processes of alpha-synucleinopathy from the prodromal phase. Indeed, identifying phenotype clusters with both consolidated and innovative biomarkers may lay the groundwork for a reliable characterization of iRBD patients, likely providing the basis for an efficient stratification of patients longitudinally followed.

Several disease-modifying therapies are now in development, including but not limited to monoclonal antibodies against alpha-synucleinopathy. Prodromal synucleinopathy patients, such as those with iRBD, are the ideal target to test disease-modifying therapies because the neurodegeneration is still in an early stage and the likelihood to rescue both brain structures and function is higher. The last aim of the FarPResto study is to have a trial-ready cohort of iRBD patients, collected with standardized and harmonized procedures, to be enrolled in upcoming disease-modifying trials.

The FARPRESTO project is endorsed by the Italian Association of Sleep Medicine (AIMS) and by The RBD_Patients society (www.sonnomed.it)

ELIGIBILITY:
Inclusion Criteria:

* Age: major of 18 years old
* iRBD diagnosis, according to diagnostic criteria of the ICSD second and third edition

Exclusion Criteria:

* Impossibility to provide or withdraw informed consent and inability to read, write and understand the purpose and modality of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged major of 18 years old, diagnosed with iRBD, that can provide informed consent referring to centers participating in the FARPRESTO study
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2035-01-31 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive risk factors of phenoconversion in patients with iRBD | May 25, 2020 - January 31, 2035
  In order to increase our understanding on the physiopathological processes of alpha-synucleinopathy from the prodromal phase clinical, biological, neurophysiological, neuropsychological and imaging biomarkers need to be prospectively collected, according to standardized and harmonized procedures. Moreover, identifying phenotype clusters with both consolidated and innovative biomakers may lay the groundwork for a reliable characterization of iRBD patients, likely providing the basis for an efficient stratification of patients to be longitudinally followed.

SECONDARY OUTCOMES:
Description of the socio-demographic and clinical characteristics of patients diagnosed with iRBD | May 25, 2020 - January 31, 2035
  Data on socio-demographic and clinical characteristics of patients diagnosed with iRBD will be collected and analyzed.
Collection of longitudinal data about the development of alpha-synucleinopathies and estimation of the conversion rate at 3, 5, 7, and 10 years | May 25, 2020 - January 31, 2035
  Information about the conversion rate at 3, 5, 7, and 10 years to neurodegenerative pathologies of the spectrum of alpha-synucleinopathies (Parkinson's Disease, Multiple System Atrophy and Lewy Body Dementia) will be collected and evaluated.
Evaluation of the impact of iRBD on the quality of life and sleep | May 25, 2020 - January 31, 2035
  The impact of iRBD on the quality of life and sleep will be assessed through the administration of validated questionnaires.
Assessment of the correlation between phenoconversion, cognitive performance and loss of normal muscle atony during REM sleep | May 25, 2020 - January 31, 2035
  The results of cognitive performance tests, video-polysomnographic recording and their connection with phenoconversion will be investigated
Identification of RBD phenotypes through different biomarkers | May 25, 2020 - January 31, 2035
  RBD phenotypes will be identified evaluating clinical, biological,neurophysiological, neuropsychological and imaging biomarkers.
Validation of vPSG criteria for RBD diagnosis | May 25, 2020 - January 31, 2035
  vPSG criteria for RBD diagnosis will be validated

CONTACTS AND LOCATIONS:
Overall Officials: Monica Puligheddu, MD,PhD, Principal Investigator — University of Cagliari
Locations (2):
- Italy (2):
  - IRCCS Auxologico Piancavallo, Oggebbio, Verbania
  - Centro Interdipartimentale di Medicina del Sonno, Università degli studi di Cagliari, Cagliari

REFERENCES:
- [Background] Fantini ML, Corona A, Clerici S, Ferini-Strambi L. Aggressive dream content without daytime aggressiveness in REM sleep behavior disorder. Neurology. 2005 Oct 11;65(7):1010-5. doi: 10.1212/01.wnl.0000179346.39655.e0. PMID 16217051
- [Background] Oudiette D, De Cock VC, Lavault S, Leu S, Vidailhet M, Arnulf I. Nonviolent elaborate behaviors may also occur in REM sleep behavior disorder. Neurology. 2009 Feb 10;72(6):551-7. doi: 10.1212/01.wnl.0000341936.78678.3a. PMID 19204265
- [Background] Schenck CH, Mahowald MW. REM sleep behavior disorder: clinical, developmental, and neuroscience perspectives 16 years after its formal identification in SLEEP. Sleep. 2002 Mar 15;25(2):120-38. doi: 10.1093/sleep/25.2.120. No abstract available. PMID 11902423
- [Background] Frauscher B, Iranzo A, Gaig C, Gschliesser V, Guaita M, Raffelseder V, Ehrmann L, Sola N, Salamero M, Tolosa E, Poewe W, Santamaria J, Hogl B; SINBAR (Sleep Innsbruck Barcelona) Group. Normative EMG values during REM sleep for the diagnosis of REM sleep behavior disorder. Sleep. 2012 Jun 1;35(6):835-47. doi: 10.5665/sleep.1886. PMID 22654203
- [Background] Anang JB, Gagnon JF, Bertrand JA, Romenets SR, Latreille V, Panisset M, Montplaisir J, Postuma RB. Predictors of dementia in Parkinson disease: a prospective cohort study. Neurology. 2014 Sep 30;83(14):1253-60. doi: 10.1212/WNL.0000000000000842. Epub 2014 Aug 29. PMID 25171928
- [Background] Anang JB, Nomura T, Romenets SR, Nakashima K, Gagnon JF, Postuma RB. Dementia Predictors in Parkinson Disease: A Validation Study. J Parkinsons Dis. 2017;7(1):159-162. doi: 10.3233/JPD-160925. PMID 27911340
- [Background] Sinforiani E, Pacchetti C, Zangaglia R, Pasotti C, Manni R, Nappi G. REM behavior disorder, hallucinations and cognitive impairment in Parkinson's disease: a two-year follow up. Mov Disord. 2008 Jul 30;23(10):1441-5. doi: 10.1002/mds.22126. PMID 18512749
- [Background] Postuma RB, Gagnon JF, Vendette M, Charland K, Montplaisir J. Manifestations of Parkinson disease differ in association with REM sleep behavior disorder. Mov Disord. 2008 Sep 15;23(12):1665-72. doi: 10.1002/mds.22099. PMID 18709686
- [Background] Postuma RB, Gagnon JF, Bertrand JA, Genier Marchand D, Montplaisir JY. Parkinson risk in idiopathic REM sleep behavior disorder: preparing for neuroprotective trials. Neurology. 2015 Mar 17;84(11):1104-13. doi: 10.1212/WNL.0000000000001364. Epub 2015 Feb 13. PMID 25681454
- [Background] Fereshtehnejad SM, Romenets SR, Anang JB, Latreille V, Gagnon JF, Postuma RB. New Clinical Subtypes of Parkinson Disease and Their Longitudinal Progression: A Prospective Cohort Comparison With Other Phenotypes. JAMA Neurol. 2015 Aug;72(8):863-73. doi: 10.1001/jamaneurol.2015.0703. PMID 26076039
- [Background] Postuma RB, Adler CH, Dugger BN, Hentz JG, Shill HA, Driver-Dunckley E, Sabbagh MN, Jacobson SA, Belden CM, Sue LI, Serrano G, Beach TG. REM sleep behavior disorder and neuropathology in Parkinson's disease. Mov Disord. 2015 Sep;30(10):1413-7. doi: 10.1002/mds.26347. Epub 2015 Aug 12. PMID 26265105
- [Background] Schenck CH, Boeve BF, Mahowald MW. Delayed emergence of a parkinsonian disorder or dementia in 81% of older men initially diagnosed with idiopathic rapid eye movement sleep behavior disorder: a 16-year update on a previously reported series. Sleep Med. 2013 Aug;14(8):744-8. doi: 10.1016/j.sleep.2012.10.009. Epub 2013 Jan 22. PMID 23347909
- [Background] Iranzo A, Fernandez-Arcos A, Tolosa E, Serradell M, Molinuevo JL, Valldeoriola F, Gelpi E, Vilaseca I, Sanchez-Valle R, Llado A, Gaig C, Santamaria J. Neurodegenerative disorder risk in idiopathic REM sleep behavior disorder: study in 174 patients. PLoS One. 2014 Feb 26;9(2):e89741. doi: 10.1371/journal.pone.0089741. eCollection 2014. PMID 24587002
- [Background] Postuma RB. Prodromal Parkinson's disease--using REM sleep behavior disorder as a window. Parkinsonism Relat Disord. 2014 Jan;20 Suppl 1:S1-4. doi: 10.1016/S1353-8020(13)00400-8. PMID 24262156
- [Background] Postuma RB, Iranzo A, Hogl B, Arnulf I, Ferini-Strambi L, Manni R, Miyamoto T, Oertel W, Dauvilliers Y, Ju YE, Puligheddu M, Sonka K, Pelletier A, Santamaria J, Frauscher B, Leu-Semenescu S, Zucconi M, Terzaghi M, Miyamoto M, Unger MM, Carlander B, Fantini ML, Montplaisir JY. Risk factors for neurodegeneration in idiopathic rapid eye movement sleep behavior disorder: a multicenter study. Ann Neurol. 2015 May;77(5):830-9. doi: 10.1002/ana.24385. Epub 2015 Mar 13. PMID 25767079
- [Background] Terzaghi M, Toscano G, Casoni F, Picascia M, Arnaldi D, Rustioni V, Versino M, Sinforiani E, Manni R. Assessment of cognitive profile as a prodromal marker of the evolution of rapid eye movement sleep behavior disorder. Sleep. 2019 Aug 1;42(8):zsz103. doi: 10.1093/sleep/zsz103. PMID 31013340
- [Background] Postuma RB, Iranzo A, Hu M, Hogl B, Boeve BF, Manni R, Oertel WH, Arnulf I, Ferini-Strambi L, Puligheddu M, Antelmi E, Cochen De Cock V, Arnaldi D, Mollenhauer B, Videnovic A, Sonka K, Jung KY, Kunz D, Dauvilliers Y, Provini F, Lewis SJ, Buskova J, Pavlova M, Heidbreder A, Montplaisir JY, Santamaria J, Barber TR, Stefani A, St Louis EK, Terzaghi M, Janzen A, Leu-Semenescu S, Plazzi G, Nobili F, Sixel-Doering F, Dusek P, Bes F, Cortelli P, Ehgoetz Martens K, Gagnon JF, Gaig C, Zucconi M, Trenkwalder C, Gan-Or Z, Lo C, Rolinski M, Mahlknecht P, Holzknecht E, Boeve AR, Teigen LN, Toscano G, Mayer G, Morbelli S, Dawson B, Pelletier A. Risk and predictors of dementia and parkinsonism in idiopathic REM sleep behaviour disorder: a multicentre study. Brain. 2019 Mar 1;142(3):744-759. doi: 10.1093/brain/awz030. PMID 30789229
- [Background] Postuma RB, Gagnon JF, Rompre S, Montplaisir JY. Severity of REM atonia loss in idiopathic REM sleep behavior disorder predicts Parkinson disease. Neurology. 2010 Jan 19;74(3):239-44. doi: 10.1212/WNL.0b013e3181ca0166. PMID 20083800
- [Background] Park JC, Moura AL, Raza AS, Rhee DW, Kardon RH, Hood DC. Toward a clinical protocol for assessing rod, cone, and melanopsin contributions to the human pupil response. Invest Ophthalmol Vis Sci. 2011 Aug 22;52(9):6624-35. doi: 10.1167/iovs.11-7586. PMID 21743008
- [Derived] Puligheddu M, Figorilli M, Antelmi E, Arnaldi D, Casaglia E, d'Aloja E, Ferini-Strambi L, Ferri R, Gigli GL, Ingravallo F, Maestri M, Terzaghi M, Plazzi G; and the FARPRESTO Consortium. Predictive risk factors of phenoconversion in idiopathic REM sleep behavior disorder: the Italian study "FARPRESTO". Neurol Sci. 2022 Dec;43(12):6919-6928. doi: 10.1007/s10072-022-06374-4. Epub 2022 Sep 10. PMID 36087148